CLINICAL TRIAL: NCT02668497
Title: Kinematic Characterization of Upper Limb Parkinson's Disease Tremor for Optimized Botulinum Toxin Type A Therapy
Brief Title: Kinematic-based BoNT-A Bilateral Upper Limb PD Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Principal Investigator, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107433
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Parkinson's Disease
Keywords: Movement disorders; Botulinum toxin type A; Tremor; Kinematics
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Tremor | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- De-novo PD (Experimental): A serotype of botulinum toxin type A (BoNT-A) that has specificity for cleavage of SYNAPTOSOMAL-ASSOCIATED PROTEIN 25 (SNAP-25). BoNT-A's pharmacological action is to inhibit the release of acetylcholine from the neuromuscular junction. BoNT-A peripherally applied using optimal parameters by intramuscular injections solely determined by biomechanical analysis of tremulous movements for tremor therapy in both upper extremity every 12 weeks over 42 weeks. BoNT-A dose will range from 50-300 U per arm
  Interventions: Drug: Botulinum Toxin Type A
- L-dopa PD (Experimental): A serotype of botulinum toxin type A (BoNT-A) that has specificity for cleavage of SYNAPTOSOMAL-ASSOCIATED PROTEIN 25 (SNAP-25). BoNT-A's pharmacological action is to inhibit the release of acetylcholine from the neuromuscular junction. BoNT-A peripherally applied using optimal parameters by intramuscular injections solely determined by biomechanical analysis of tremulous movements for tremor therapy in both upper extremity every 12 weeks over 42 weeks. BoNT-A dose will range from 50-300 U per arm
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Other Names: IncobotulinumtoxinA; BoNT-A

SUMMARY:
The primary objective is to study the efficacy of botulinum toxin type A (BoNT-A) injected via kinematic parameters in the treatment of unilateral/bilateral upper extremity tremor in Parkinson's disease (PD) tremor. Kinematic assessment tools already developed in past clinical studies will be used in determining injection parameters. The objective is to study the composition of PD tremor using kinematic tools which may contribute to the knowledge of tremor complexity and contribute information that would benefit the development of injection parameters to improve efficacy and optimization of BoNT-A in tremor management. By injecting all bothersome tremulous upper limbs in Parkinson's disease patients, the investigators believe a greater improvement in Quality of Life on more daily tasks can be achieved compared to the investigator's earlier study in unilateral injections (REB#101749), which already showed significant improvement.

ELIGIBILITY:
Inclusion Criteria:

* PD individuals diagnosed by UK Brain Bank Criteria with stage H&Y2-3 disease
* PD participants who are naïve to PD medications will be grouped into the "De novo" PD group
* PD participants stable on a low dose of Levodopa or on their PD medications for at least 3 months prior to their study enrolment will be grouped into the "L-dopa" PD group
* Participants who are botulinum toxin naïve for tremor management
* Patients will be screened for pregnancy by the physician
* Individuals with PD will be eligible for the study only if tremor is their primary and most bothersome symptom as determined by clinical exam and patient report denoting tremor-dominant phenotype
* Participants must be able to provide informed consent and to complete all study assessment scales and tasks.

Exclusion Criteria:

* History of stroke
* History of ALS or Myasthenia Gravis
* History of COPD or emphysema
* Underlying arm muscle weakness or any related compartmental muscle syndrome
* Offending medications (Lithium, valproate, steroids, amiodarone, beta-adrenergic agonists (e.g. salbutamol).
* Persons prescribed zonisamide
* History of allergic or side effect reaction to botulinum toxin
* Contraindications per the BoNT-A drug monograph
* Women reporting that they are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Kinematic tremor severity | 42 weeks
  Change from pre to post-BoNT-A treatments in maximum angular tremor amplitude at the wrist in each treated arm. Angular tremor amplitude is one parameter reflecting the vectoral intensity of tremor segmented at each arm joint

SECONDARY OUTCOMES:
Clinical tremor severity | 42 weeks
  Improvement in upper limb tremor severity as determined by an increase >8 points on a standardized clinical assessment tool (Fahn-Tolosa-Marin Tremor Assessment Scale) pre and post BoNT-A injection using kinematic-determined injection parameters in both ET upper limbs
Accelerometric kinematic tremor severity | 42 weeks
  Change from pre and post-BoNT-A treatments in maximum log-transformed accelerometric tremor amplitude at wrist level (injected limb). Log-transformed accelerometric tremor amplitude is one parameter reflecting the non-vectoral intensity of tremor.
Quality of life measures | 42 weeks
  Quality of life for essential tremor questionnaire is used to measure the patient's impression of change due to treatment and its change on their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — LHSC
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Milanov I. A cross-over clinical and electromyographic assessment of treatment for parkinsonian tremor. Parkinsonism Relat Disord. 2001 Sep;8(1):67-73. doi: 10.1016/s1353-8020(00)00077-8. PMID 11472883
- [Background] Kraus PH, Lemke MR, Reichmann H. Kinetic tremor in Parkinson's disease--an underrated symptom. J Neural Transm (Vienna). 2006 Jul;113(7):845-53. doi: 10.1007/s00702-005-0354-9. Epub 2006 Jan 30. PMID 16804646
- [Background] Jimenez MC, Vingerhoets FJ. Tremor revisited: treatment of PD tremor. Parkinsonism Relat Disord. 2012 Jan;18 Suppl 1:S93-5. doi: 10.1016/S1353-8020(11)70030-X. PMID 22166467
- [Background] Imbach LL, Sommerauer M, Leuenberger K, Schreglmann SR, Maier O, Uhl M, Gassert R, Baumann CR. Dopamine-responsive pattern in tremor patients. Parkinsonism Relat Disord. 2014 Nov;20(11):1283-6. doi: 10.1016/j.parkreldis.2014.09.007. Epub 2014 Sep 16. PMID 25260965
- [Background] Miyasaki JM, Martin W, Suchowersky O, Weiner WJ, Lang AE. Practice parameter: initiation of treatment for Parkinson's disease: an evidence-based review [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2002 Jan 8;58(1):11-7. doi: 10.1212/wnl.58.1.11. PMID 11781398
- [Background] Nagatsua T, Sawadab M. L-dopa therapy for Parkinson's disease: past, present, and future. Parkinsonism Relat Disord. 2009 Jan;15 Suppl 1:S3-8. doi: 10.1016/S1353-8020(09)70004-5. PMID 19131039
- [Background] Stathis P, Konitsiotis S, Antonini A. Dopamine agonists early monotherapy for the delay of development of levodopa-induced dyskinesias. Expert Rev Neurother. 2015 Feb;15(2):207-13. doi: 10.1586/14737175.2015.1001747. Epub 2015 Jan 12. PMID 25578445
- [Background] Katzenschlager R, Sampaio C, Costa J, Lees A. Anticholinergics for symptomatic management of Parkinson's disease. Cochrane Database Syst Rev. 2003;2002(2):CD003735. doi: 10.1002/14651858.CD003735. PMID 12804486